CLINICAL TRIAL: NCT02157727
Title: Effectiveness and Cost-effectiveness of Tele-expertise for the Screening Examination of Premature Infants for Retinopathy of Prematurity
Brief Title: Cost-effectiveness of Tele-expertise for Premature Infants for Retinopathy
Acronym: Dite-ROP
Status: Completed | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: Agence Regionale de Sante d'Ile de France (Other Government)
Responsible Party: Sponsor
Other Study IDs: TLM-DITEROP
Record Dates: First submitted 2014-05-27; First posted 2014-06-06 (Estimated); Last update posted 2015-10-14 (Estimated); Status verified 2015-10

CONDITIONS: Retinopathy of Prematurity
MeSH Terms: conditions — Retinopathy of Prematurity

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- Exposed group, during Tele-expertise: Infants hospitalized in health facilities performing tele-expertise
  Interventions: Device: Infants hospitalized in health facilities performing Tele-expertise
- Exposed group, Prior Tele-expertise: Infants hospitalized in health facilities performing Tele-expertise prior implementation of Tele-expertise
- Control group, Prior Tele-expertise
- Control group, during Tele-expertise: Infants hospitalized in health facilities not performing Tele-expertise while the exposed group use Tele-expertise

INTERVENTIONS:
Device: Infants hospitalized in health facilities performing Tele-expertise
  Groups: Exposed group, during Tele-expertise

SUMMARY:
The purpose of this study is to determine whether telemedicine would be as effective as having a pediatrics ophthalmologist on site for screening examination of retinopathy in premature infants and would be cost-effective.

ELIGIBILITY:
Inclusion Criteria:

* Born before 32 WA or having a birth weight under 1500g

Exclusion Criteria:

* Brain malformations

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Infants hospitalized in neonatology unit
Sampling Method: Non-Probability Sample
Enrollment: 843 (Actual)
Dates: Start 2014-01; Primary Completion 2015-06 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Proportion of premature infants being screened for retinopathy following recommendations | 4 weeks in average
  Proportion of premature infants being screened for retinopathy following recommendations (between 31 and 32 weeks of amenorrhea (WA) for infants born before 28 WA and during the fourth week of life for infants born after 28 WA)

SECONDARY OUTCOMES:
Delay before the first screening of retinopathy | 4 weeks in average
  For infants born at or after 28WA
Cost of telemedicine | 6 months after enrollment of the first patient

CONTACTS AND LOCATIONS:
Overall Officials: Isabelle Durand-Zaleski, MD, PhD, Principal Investigator — DRCD URC Eco. Assistance Publique, Hôpitaux de Paris; Michele Granier, MD, Principal Investigator — Centre Hospitalier Sud Francilien
Locations (2):
- France (2):
  - Service de réanimation néonatale. Centre Hospitalier Sud Francilien, Corbeil-Essonnes
  - Service de réanimation néonatale. Maternité de Port-Royal, Paris

REFERENCES:
- [Background] Kidholm K, Ekeland AG, Jensen LK, Rasmussen J, Pedersen CD, Bowes A, Flottorp SA, Bech M. A model for assessment of telemedicine applications: mast. Int J Technol Assess Health Care. 2012 Jan;28(1):44-51. doi: 10.1017/S0266462311000638. PMID 22617736
- [Background] Fierson WM; American Academy of Pediatrics Section on Ophthalmology; American Academy of Ophthalmology; American Association for Pediatric Ophthalmology and Strabismus; American Association of Certified Orthoptists. Screening examination of premature infants for retinopathy of prematurity. Pediatrics. 2013 Jan;131(1):189-95. doi: 10.1542/peds.2012-2996. Epub 2012 Dec 31. PMID 23277315
- [Derived] Charrier N, Zarca K, Durand-Zaleski I, Calinaud C; ARS Ile de France telemedicine group. Efficacy and cost effectiveness of telemedicine for improving access to care in the Paris region: study protocols for eight trials. BMC Health Serv Res. 2016 Feb 8;16:45. doi: 10.1186/s12913-016-1281-1. PMID 26857558